CLINICAL TRIAL: NCT00900783
Title: A Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Comparative Study of FV-100 vs. Valacyclovir in Patients With Herpes Zoster
Brief Title: A Study of FV-100 Versus Valacyclovir in Patients With Herpes Zoster
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INH-FV1-005; INH-FV1-005-PK; INH-FV1-005-VR; INH-FV1-AGE
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Herpes Zoster; Shingles
Keywords: herpes zoster; shingles; Phase II; FV-100; Inhibitex
MeSH Terms: conditions — Herpes Zoster | interventions — Valacyclovir; FV-100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Experimental): FV-100, 400 mg once daily AND valacyclovir placebo, three times a day, for seven days
  Interventions: Drug: FV-100; Drug: Valacyclovir placebo
- 3 (Active Comparator): Valacyclovir, 1 gram, three times a day AND FV-100 placebo, once daily, for seven days
  Interventions: Drug: valacyclovir; Drug: FV-100 placebo
- 1 (Experimental): FV-100, 200 mg once daily AND valacyclovir placebo, three times a day, for seven days
  Interventions: Drug: FV-100; Drug: Valacyclovir placebo

INTERVENTIONS:
Drug: valacyclovir — 1 gram, three times a day for seven days
  Other Names: Valtrex
  Arms: 3
Drug: FV-100 — 400 mg, once daily, for seven days
  Arms: 2
Drug: FV-100 — 200 mg, once daily, for seven days
  Arms: 1
Drug: Valacyclovir placebo — three times a day, for seven days
  Arms: 1; 2
Drug: FV-100 placebo — once daily, for seven days
  Arms: 3

SUMMARY:
The purpose of this study is to compare the safety and efficacy of two doses of FV-100 to valacyclovir in patients with herpes zoster, or shingles. FV-100 has shown to be very potent in cells infected with varicella zoster virus, the virus that causes shingles. The study objectives include:

* Compare the safety of FV-100 to valacyclovir
* Compare the effect of FV-100, as compared to valacyclovir, on shingles pain
* Compare the effect of FV-100, as compared to valacyclovir, on shingles lesions

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years of age
* Patients with a clinical diagnosis of HZ as evidenced by a unilateral dermatomal rash
* Patients with zoster-related pain (ZBPI worst pain score > 0)
* Patients able to be enrolled into the study ≤ 72 hours from appearance of rash (i.e., lesions or vesicles)
* Patients providing written informed consent
* Patients who are able to complete all study visits per protocol
* Men and premenopausal women must agree to practice a barrier method of birth control plus the use of a spermicide for one month after the last dose of study drug (oral contraceptives are not permitted)

Exclusion Criteria:

* Women who are pregnant or lactating
* Patients with multidermatomal or disseminated HZ (i.e., > 20 vesicles beyond the dermatomes adjacent to the primarily involved dermatome)
* Patients with HZ ophthalmicus, defined as cutaneous lesions in the dermatome associated with the ophthalmic division of the trigeminal nerve
* Patients with history of impaired renal function, (e.g., calculated creatinine clearance <50 mL/min/1.73 m2)
* Patients taking narcotic analgesic routinely for a chronic pain condition
* Patients taking tricyclic antidepressants
* Patients who have received systemic antivirals with activity against VZV within the past 30 days, or a topical antiviral to treat their current HZ
* Patients who are immunosuppressed from:

  * disease (e.g., malignancy [present or remission < 5 years], HIV)
  * corticosteroid use (except intermittent or topical/inhaled beclomethasone dipropionate or equivalent < 800 mcg/day), or
  * other immunosuppressive/cytotoxic therapy (cancer chemotherapy or organ transplantation)
* Patients with gastrointestinal dysfunction that could interfere with drug absorption
* Patients with any other condition (e.g., extensive psoriasis, chronic pain syndrome, cognitive impairment) that, in the opinion of the site investigator, might interfere with the evaluations required by the study
* Patients who are not ambulatory (bed-ridden or homebound); hospitalized patients may be enrolled if they are ambulatory and able to complete the study requirements
* Patients with history of allergy to valacyclovir hydrochloride
* Patients unlikely to adhere to protocol follow-up
* 14. Subjects taking strong CYP3A4-inhibiting protease inhibitors (specifically including atazanavir, indinavir, nelfinavir, saquinavir, and ritonavir), strong CYP3A4 inhibitors (specifically including clarithromycin, itraconazole, ketoconazole, nefazodone, telithromycin) and all strong CYP3A4 inducers (specifically including rifampin, efavirenz, etravirine, phenobarbital, phenytoin, and carbamazepine)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Herpes zoster associated pain, as measured by the Zoster Brief Pain INventory (ZBPI) | 30 days

SECONDARY OUTCOMES:
Herpes zoster associated pain | 90 days
Herpes zoster lesion healing | Until healed
Routine clinical labs | 30 days

REFERENCES:
- [Derived] Tyring SK, Lee P, Hill GT Jr, Silverfield JC, Moore AY, Matkovits T, Sullivan-Bolyai J. FV-100 versus valacyclovir for the prevention of post-herpetic neuralgia and the treatment of acute herpes zoster-associated pain: A randomized-controlled trial. J Med Virol. 2017 Jul;89(7):1255-1264. doi: 10.1002/jmv.24750. Epub 2016 Dec 26. PMID 27943311